CLINICAL TRIAL: NCT05834088
Title: Effects of Myofascial Release With and Without Thiele Massage on Dyspareunia and Pelvic Floor Function in Nulliparous Females
Brief Title: Effects of Myofascial Release With and Without Thiele Massage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0513
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Dyspareunia; Pain; Quality of Life
Keywords: Dyspareunia; Pelvic floor disorder; Pelvic pain; Myofascial release technique; Pelvic floor
MeSH Terms: conditions — Dyspareunia; Pain; Pelvic Floor Disorders; Pelvic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial techniques with Thiele massage (Experimental): Group A will receive myofascial techniques with Thiele massage. 12 treatment sessions will be given in 12 weeks
  Interventions: Other: Myofascial release techniques; Other: Thiele massage
- Myofascial techniques without Thiele massage (Active Comparator): Group B will receive myofascial techniques without Thiele massage. 12 treatment sessions will be given in 12 weeks
  Interventions: Other: Myofascial release techniques

INTERVENTIONS:
Other: Myofascial release techniques — 12 treatment sessions will be given in 12 weeks
Other: Thiele massage — 12 treatment sessions will be given in 12 weeks
  Arms: Myofascial techniques with Thiele massage

SUMMARY:
Dysperunia is caused by chronic discomfort during sexual intercourse causing pain during vaginal intercourse.Sexual pain causes relationship decreasing quality of life following anxiety and depression.Myofascial techniques with and without Thiele massage will be used via randomised controlled trial following sample size of 38.

DETAILED DESCRIPTION:
Dyspareunia is characterised by recurring or chronic discomfort during sexual intercourse that causes distress. Dyspareunia can be superficial, causing pain when vaginal insertion is tried, or profound. Women who experience sexual pain are more likely to experience sexual dysfunction, relationship distress, decreased quality of life, anxiety, and depression. One in five nulliparous women (a female who has never given birth to a baby) experiences moderate dyspareunia. Myofascial pain is typically treated using manual manipulation (Manual manipulation involves using skilled, hands-on maneuvers to perform soft tissue mobilization, myofascial release and more) or Thiele massage. In this study the aim is to find the individual and combined effect of these techniques. The study will be Randomized Controlled Trial (RCT). Non probabiity convenient sampling technique will be used to assign randomly half of patients in group A for the experimental group and half in group B who will meet the inclusion criteria. Group A will include participants who will receive myofascial releases and Thiele massage. Whereas Group B will include participants who will receive myofascial releasing techniques but not Thiele massage.

Both group will have 1 session per week for 12 weeks. Numeric pain rating scale, Female sexual function index, Functional pelvic pain scale would be used as an outcome measure tools.

The collected data will be analyzed in Statistical Package for the Social Sciences (SPSS) 25

ELIGIBILITY:
Inclusion Criteria:

Age 23-40

1. Dyspareunia symptoms for more than 6 months
2. Females with tenderness of pelvic muscles from last 6 months
3. Nulliparous women

Exclusion Criteria:

1. Any pelvic organ prolapse
2. Any current genital malignancy
3. Cases of chronic pelvic pain due to any other issue
4. Any traumatic conditions around the pelvis and lower limbs, any infectious, tumors conditions around the pelvis.
5. Pregnant females
6. Any lower limb abnormalities, any recently underwent abdominal and low back surgery.

Ages: 23 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Nulliparous females
Enrollment: 38 (Actual)
Dates: Start 2022-11-20 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale | 12 weeks
  The numeric rating scale (NRS) is a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable".
Female sexual function index | 12 weeks
  The FSFI is a widely-used measure of Female Sexual Dysfunction (FSD). It assesses 6 domains: desire; arousal; lubrication; orgasm; satisfaction; and pain.
Functional pelvic pain scale | 12 weeks
  Functional Pelvic Pain Scale (FPPS), designed to measure pelvic pain intensity as it relates to functions of daily living (bladder and bowel function, intercourse, walking, running, lifting, working, and sleeping).

CONTACTS AND LOCATIONS:
Overall Officials: Sabiha Arshad, M.phil, Principal Investigator — Riphah International University
Locations (1):
- Jinnah hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mitchell KR, Geary R, Graham CA, Datta J, Wellings K, Sonnenberg P, Field N, Nunns D, Bancroft J, Jones KG, Johnson AM, Mercer CH. Painful sex (dyspareunia) in women: prevalence and associated factors in a British population probability survey. BJOG. 2017 Oct;124(11):1689-1697. doi: 10.1111/1471-0528.14518. Epub 2017 Jan 25. PMID 28120373
- [Background] Tayyeb M, Gupta V. Dyspareunia. 2023 Jun 5. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK562159/ PMID 32965830
- [Background] Castellanos-Lopez E, Castillo-Merino C, Abuin-Porras V, Lopez-Lopez D, Romero-Morales C. Ultrasonography Comparison of Pelvic Floor and Abdominal Wall Muscles in Women with and without Dyspareunia: A Cross-Sectional Study. Diagnostics (Basel). 2022 Jul 29;12(8):1827. doi: 10.3390/diagnostics12081827. PMID 36010178
- [Background] Rosen NO, Dawson SJ, Binik YM, Pierce M, Brooks M, Pukall C, Chorney J, Snelgrove-Clarke E, George R. Trajectories of Dyspareunia From Pregnancy to 24 Months Postpartum. Obstet Gynecol. 2022 Mar 1;139(3):391-399. doi: 10.1097/AOG.0000000000004662. PMID 35115480
- [Background] Alimi Y, Iwanaga J, Oskouian RJ, Loukas M, Tubbs RS. The clinical anatomy of dyspareunia: A review. Clin Anat. 2018 Oct;31(7):1013-1017. doi: 10.1002/ca.23250. Epub 2018 Oct 26. PMID 30113086
- [Background] Geller EJ, Babb E, Nackley AG, Zolnoun D. Incidence and Risk Factors for Pelvic Pain After Mesh Implant Surgery for the Treatment of Pelvic Floor Disorders. J Minim Invasive Gynecol. 2017 Jan 1;24(1):67-73. doi: 10.1016/j.jmig.2016.10.001. Epub 2016 Oct 20. PMID 27773810